CLINICAL TRIAL: NCT05873582
Title: Robotic Minimally Invasive Inguinal Hernia Repair With Dexter
Acronym: RAS-Ahead
Status: Completed | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-01
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Inguinal Hernia Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Robotic-assisted inguinal hernia repair — Primary transperitoneal unilateral or bilateral inguinal hernia repair with the Dexter robotic system

SUMMARY:
This study aims to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing primary transperitoneal unilateral or bilateral inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patients planned to undergo elective robot-assisted and laparoscopic surgery for primary unilateral or bilateral inguinal hernia repair using one camera port, two ports for the manipulating instruments, and additional ports as needed.
* Able to provide Informed Consent according to local regulation

Exclusion Criteria:

* Morbidly obese patients (BMI > 40)
* Any relative and absolute contraindications for the use of conventional endoscopes and endoscopic surgical instruments
* Need for robotic stapling, advanced energy delivery, ultrasound, cryoablation and microwave energy delivery
* Bleeding diathesis
* Pregnancy
* Patients with pacemakers or internal defibrillators
* Any planned concomitant procedures
* Patient deprived of liberty by administrative or judicial decision or under legal guardianship
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing primary transperitoneal unilateral or bilateral inguinal hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Safety: occurrence of serious (Clavien - Dindo grades III-V), device-related, adverse events | perioperatively up to 30 days
Performance: successful completion of the Dexter-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach | intraoperative

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Hospitalier de Saintes, Saintes, France
- UKSH Kiel, Kiel, Germany
- Kantonspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: No